CLINICAL TRIAL: NCT02785679
Title: The Influence of Early and Continuous Exposure of Infants to Cow's Milk Formula on the Prevention of Milk Allergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Schneider Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 011-16-MMC
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Cow Milk Allergy; Newborns
Keywords: Allergy; Cow's milk; breast feeding; Cow's milk formula; prevention
MeSH Terms: conditions — Milk Hypersensitivity; Hypersensitivity; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exclusive breast feeding (No Intervention): Exclusive breast feeding
- Exclusive CMF feeding (No Intervention): Exclusive CMF feeding
- Breast feeding with small amount of CMF (Active Comparator): Breast feeding with addition (as intervention) of 20 cc of cow's milk formula (CMF) per day
  Interventions: Dietary Supplement: cow's milk formula
- Breast feeding with one meal of CMF (Active Comparator): Breast feeding with addition (as intervention) of one meal per day of cow's milk formula (CMF)
  Interventions: Dietary Supplement: cow's milk formula

INTERVENTIONS:
Dietary Supplement: cow's milk formula — addition of cow's milk formula in two different dosage - one only 20ml per day and one group a full meal per day
  Arms: Breast feeding with one meal of CMF; Breast feeding with small amount of CMF

SUMMARY:
Cow's milk protein (CMP) allergy is one of the most common food allergies and potentially a fatal one. Early feeding with CMP has been considered in the past as a risk factor for development of CMP allergy in high risk infants. Although other studies argue with this assumption and suggest early exposure to CMP might be protective against atopic dermatitis and CMP allergy. A cohort study that first introduction of CMP after 15-30 days of age, raised the risk for CMP allergy.The aim of this study is to investigate if early and continuous exposure to CMF will decrease CMP allergy rate.

DETAILED DESCRIPTION:
Background: Cow's milk protein (CMP) allergy is one of the most common food allergies and potentially a fatal one. The incidence of milk allergy is 1.5-3% in the first year of life, but only 60% of the reactions are IgE mediated. CMP allergy tends to resolve in approximately 45-50% of the infants at 1 year of age, in 60-75% at the age of 2, and 85-90% at 3 years. The range for IgE mediated CMP allergy is 29-76%. A recent study suggested that the natural history of CMP allergy might have changed over time, with slower rates of resolution and a higher proportion of children with disease persisting into adolescence and adulthood. In the past it has been described that there is more incidence of CMP allergy in children from families with positive history of allergy. Early feeding with CMP has been considered in the past as a risk factor for development of CMP allergy in high risk infants. Although other studies argue with this assumption and suggest early exposure to CMP might be protective against atopic dermatitis and CMP allergy. A cohort study that first introduction of CMP after 15-30 days of age, raised the risk for CMP allergy. A recent study on peanut allergy found that continuous early exposure to peanut dramatically decreased the incidence of peanut allergy. The research in the field of food allergy and especially in CMP allergy is very alert those days. But as far as the investigators knowledge, there are no prospective studies from the first days of life that examined the influence of early and continuous exposure to cow's milk formula (CMF) on CMP allergy. The existing data related to CMP allergy is controversial and inconclusive. Thus, no one can rely on it to establish clear recommendations for parents when is the best time to combine CMF in the infants diet. Working hypothesis and aims: The aim of the study is to investigate if early and continuous exposure to CMF will decrease CMP allergy rate. The investigators assumption is that the rate of CMP allergy in the intervention groups and in infants who are only feed by CMF, will be lower than in the group of infants who are exclusively breast feed. Methods: Recruitment of 2,500 infants from first day of life and divide the participants into 4 groups: 1. Exclusive breast feeding. 2. Exclusive CMF feeding. 3. Breast feeding with 20 cc of CMF per day. 4. Breast feeding with one meal per day of CMF. The mother will complete a survey questionnaire before the labor. Infants will be followed for 1 year. During this follow-up period -the participants will be examined by an allergologist at the age of 2 month and 1 year. In between, the infants will be followed by a phone questionnaire once in a month. Specific CM IgE analysis from umbilical cord blood and skin test at 2 month of age will be performed. Inclusion criteria - Term and near term newborns (gestational age of at least 36 weeks), normal birth weight, normal perinatal follow-up and without congenital defects. Expected results: The rate of CMP allergy in the intervention groups and in the group on exclusively CMF feeding will be lower than in the group on exclusive breast feeding. Importance: If the investigators will be able to prove the study hypothesis (and even if not), it will have a significant influence on the diet recommendations for infants. Probable implications to Medicine: If the investigators will get the expected results, the recommendations that exist today for infant's feeding can be changed.

ELIGIBILITY:
Inclusion Criteria:

* Term and near term newborns (gestational age of at least 36 weeks)
* normal birth weight
* normal perinatal follow-up (physiological neonatal jaundice is not an exclusion criteria)
* without congenital defects

Exclusion Criteria:

* Preterm newborns
* Congenital defects
* Newborn suffering from acute event

Ages: 2 Hours to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2500 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of cow's milk allergy in the intervention groups | 1 year
  Measure the rate of cow's milk allergy infants in each group and compare the rate of allergy between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Confino- Cohen, MD, Study Director — allergy and immunology unit, MeirMc
Locations (1):
- Meir medical center, Kfar Saba, Israel

REFERENCES:
- [Derived] Lachover-Roth I, Cohen-Engler A, Furman Y, Rosman Y, Meir-Shafrir K, Mozer-Mandel M, Farladansky-Gershnabel S, Biron-Shental T, Confino-Cohen R. Infants born during COVID-19 pandemic experience increased susceptibility to airway hyperresponsiveness. Front Allergy. 2024 Dec 16;5:1512182. doi: 10.3389/falgy.2024.1512182. eCollection 2024. PMID 39737062
- [Derived] Lachover-Roth I, Cohen-Engler A, Furman Y, Rosman Y, Meir-Shafrir K, Mozer-Mandel M, Farladansky-Gershnabel S, Biron-Shental T, Confino-Cohen R. Food allergy and infant feeding practices: Are they related? Ann Allergy Asthma Immunol. 2023 Sep;131(3):369-375.e3. doi: 10.1016/j.anai.2023.05.031. Epub 2023 Jun 1. PMID 37270027